CLINICAL TRIAL: NCT05338749
Title: An Open-label Trial of Computer-delivered Cognitive Training in Persons With Post-acute COVID-19 Syndrome
Brief Title: Computer Cognitive Training for Post-acute COVID-19 Syndrome
Acronym: PACS-Cog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20211020
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Corona Virus Infection; Cognitive Dysfunction
MeSH Terms: conditions — Coronavirus Infections; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Training (Experimental): Participants in this condition will received game-based cognitive training.
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Gamified cognitive training intervention to improve mental speed and attention.

SUMMARY:
This study will assess the acceptability, feasibility, and impact of game-based computer-delivered cognitive training on cognitive function in persons with cognitive symptoms that persist after recovery from acute coronavirus-19 (COVID) infection.

DETAILED DESCRIPTION:
Over the course of the past several years, it has become apparent that a number of individuals have residual symptoms after COVID-19 infection after they have recovered from the acute phase of the illness (Al-Aly, Xie, & Bowe, 2021; Davis et al., 2021; Greenhalgh, Knight, A'Court, Buxton, & Husain, 2020; Hewitt et al., 2021). The constellation of symptoms experienced by these individuals has been termed "post-acute COVID syndrome" or PACS (Nalbandian et al., 2021). A key part of helping affected individuals is supporting their efforts at self-management of these symptoms (National Institute for Health and Care Excellence, 2020; Wade, 2020). Although a diverse number of physical and psychological symptoms have been seen as sequelae of COVID (Davis et al., 2021), among the most troubling for patients have been difficulties in attention, concentration, working memory, and long-term memory, commonly referred to as "brain fog" (Graham et al., 2021; Hampshire et al., 2021; Hewitt et al., 2021). In the proposed study, we will complete a pilot study of game-based cognitive training in persons with symptoms of long COVID using a protocol that was useful and acceptable to participants in a previous study (Ownby & Kim, 2021). We will explore participants' views on the cognitive training intervention, its effects on their perceived cognitive functioning, and assess the intervention's impact on participants' processing speed. We will also explore their preferences for type of cognitive training activity and the impact of information about memory functioning.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a history of COVID-19 infection confirmed through screening of symptom pattern or testing and report of mental symptoms (difficulties in attention, memory, or executive functions such as coordinating two activities at once) more than 30 days after resolution of the initial acute infection.

Exclusion Criteria:

* Cognitive or psychiatric conditions of a severity that precludes the person's ability to give informed consent for their participation or to attend and cooperate with assessment and training, as judged by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Technology Acceptance Model Questionnaire, Usefulness subscale | Three weeks
  User self-report of their perception that an application serves a function that may be helpful The score is the average of several items rated by the user from 0 to 6, so that the final score itself can range from 0 to 6. Higher scores indicate that the user found the intervention more useful. Higher scores are better.

SECONDARY OUTCOMES:
Cognitive Failures Questionnaire | Three weeks
  A standard self-report measure of problems in memory, attention, and self-regulated behavior. This measures includes self-report ratings on 25 items, with ratings ranging from 0 to 4. The total score can thus range from 0 to 100, with higher scores indicating that the person experiences more problems with thinking and remembering.
Trail Making Test, Part B | Three weeks
  This is a measure of how rapidly a person can remember alternating sequences of numbers and letters while connecting them on a paper with a pencil. The score is time in seconds to complete the task, with the provision that if a person cannot finish the task within three minutes, the task is discontinued and the person is assigned a score of 180 (for 3 minutes times 60 seconds). Lower scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Ownby, MD, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Center for Collaborative Research, Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan
Supporting Information: Study Protocol, SAP
Time Frame: After completion of study
Access Criteria: On request from any qualified investigator.

REFERENCES:
- [Background] Ownby RL, Kim J. Computer-Delivered Cognitive Training and Transcranial Direct Current Stimulation in Patients With HIV-Associated Neurocognitive Disorder: A Randomized Trial. Front Aging Neurosci. 2021 Nov 15;13:766311. doi: 10.3389/fnagi.2021.766311. eCollection 2021. PMID 34867291